CLINICAL TRIAL: NCT00115986
Title: A Randomized, Double-Blinded, Placebo-Controlled, Phase I/II, Dose-Ranging Study of the Safety, Reactogenicity, and Immunogenicity of Intramuscular Inactivated Influenza A/H5N1 Vaccine in Healthy Adults
Brief Title: A/H5N1in Adult - Aventis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04-063
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2007-01

CONDITIONS: Influenza
Keywords: A/H5N1, Influenza, Vaccine, parent protocol
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: Influenza A/H5N1 Vaccine

SUMMARY:
The purpose of this research study is to compare how the body reacts to different strengths of the new H5N1 flu vaccine. The study will also look at how antibodies are made after a subject receives the H5N1 flu vaccine. The vaccine will be given as a shot in the arm. Participants will be randomly assigned to receive 1 of 4 different dosages of the vaccine or a placebo (dummy) dose of the vaccine. Study procedures will include a physical exam, a urine pregnancy test for women, and blood samples. Participants will be asked to complete a diary to record temperatures, medications taken, and side effects from the vaccine. Volunteers will be involved with study procedures for approximately 7 months. The study will enroll about 450-470 healthy participants, ages 18-64.

DETAILED DESCRIPTION:
Approximately 450 healthy adults, 18 to 64 years old, inclusive, will be enrolled into this multicenter, randomized, double-blinded, placebo-controlled, dose-ranging clinical trial. The study will be conducted in 2 stages. During Stage I, 113 subjects who meet the entry criteria for the study will be randomized to receive saline placebo, or 7.5, 15, 45, or 90 mcg of the influenza A/H5N1 vaccine by intramuscular injection in an approximate 1:2:2:2:2 ratio (N=25/vaccine dose group and 13 in the placebo group). Subjects will receive 2 doses separated by approximately 28 days. Vaccine administration will be performed by an unblinded vaccine administrator, who will not be involved in subsequent assessments. Subjects will be observed in the clinic for 15 to 30 minutes after inoculation, and subjects will maintain a memory aid to record oral temperature and systemic and local AEs for 7 days after each immunization. Subjects will be contacted by telephone on Day 2 after each immunization to assess for the occurrence of AEs, and they will return on Day 7 for AE and concomitant medication assessment, a targeted physical examination (if indicated), and review of the memory aid. Serum for immunogenicity evaluations will be obtained prior to the first vaccination (ie, at screening for Stage I and Day 0 for Stage II), prior to the second vaccination, at Day 28, and on Days 56 and 208. All available 7-day safety data following the first dose of vaccine on the 113 subjects enrolled in Stage I will be reviewed by the Safety Monitoring Committee (SMC) prior to enrollment of the remaining subjects (Stage II), who will be followed according to the same protocol. All available 7-day safety data following the second dose of vaccine on the subjects enrolled in Stage I also will be reviewed by the SMC prior to administering the second dose of vaccine to the subjects in Stage II. This study is linked to DMID protocols 07-0022, 05-0006, 05-0090 and 08-0059.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to participate in this study: 1. Male or nonpregnant female (as indicated by a negative urine pregnancy test immediately prior to vaccine administration) between the ages of 18 and 64 years, inclusive. 2. Women of childbearing potential who are at risk of becoming pregnant must agree to practice adequate contraception (ie, barrier method, abstinence, and licensed hormonal methods) for the entire study period. 3. Is in good health, as determined by vital signs (heart rate, blood pressure, oral temperature), medical history and a targeted physical examination based on medical history. 4. In Stage I subjects, should have normal laboratory values of Hgb, WBC, Plt, ALT, and creatinine prior to the first immunization. 5. Able to understand and comply with planned study procedures. 6. Provides informed consent prior to any study procedures and is available for all study visits.

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria at baseline will be excluded from study participation: 1. Has a known allergy to eggs or other components of the vaccine. 2. Has a positive urine pregnancy test prior to vaccination (if female of childbearing potential) or women who are breastfeeding. 3. Is undergoing immunosuppression as a result of an underlying illness or treatment. 4. Has an active neoplastic disease or a history of any hematologic malignancy. 5. Is using oral or parenteral steroids, high-dose inhaled steroids (>800 µg/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs. 6. Has a history of receiving immunoglobulin or other blood product within the 3 months prior to enrollment in this study. 7. Has received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study. 8. Has an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses (this includes, but is not limited to: known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients). 9. Has a history of severe reactions following immunization with contemporary influenza virus vaccines. 10. Has an acute illness, including an oral temperature greater than 100.4ºF, within 1 week of vaccination. 11. Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to enrollment in this study, or expects to receive an experimental agent during the 7-month study period. 12. Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 452 (Actual)
Dates: Start 2005-03; Study Completion 2006-02

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UCLA Center For Vaccine Research, Torrance, California
  - University of Maryland Baltimore, Baltimore, Maryland
  - University of Rochester Medical Center - Strong Memorial Hospital - Infectious Diseases, Rochester, New York

REFERENCES:
- [Result] Treanor JJ, Campbell JD, Zangwill KM, Rowe T, Wolff M. Safety and immunogenicity of an inactivated subvirion influenza A (H5N1) vaccine. N Engl J Med. 2006 Mar 30;354(13):1343-51. doi: 10.1056/NEJMoa055778. PMID 16571878